CLINICAL TRIAL: NCT05137145
Title: Effect and Safety of Polyethylene Glycol Combined With Linaclotide on Colon Cleansing Before Colonoscopy in Patients With Chronic Constipation:an Endoscopist-blinded,Randomized,Controlled, Multicentre Trial
Brief Title: Effect and Safety of Polyethylene Glycol Combined With Linaclotide on Colon Cleansing for Patients With Chronic Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2021030
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Bowel Preparation
Keywords: Chronic Constipation; Colonoscopy; Linaclotide
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The control group (Experimental): The control group was given 4L of Compound Polyethylene Glycol Electrolyte Powder to clear the intestines
  Interventions: Drug: Compound Polyethylene Glycol Electrolyte Powder
- the observation group 1 (Experimental): the observation group 1 was given Linaclotide(290 ug) in 1 day combined with 4L of Compound Polyethylene Glycol Electrolyte Powder to clear the intestine
  Interventions: Drug: Linaclotide; Drug: Compound Polyethylene Glycol Electrolyte Powder
- the observation group 2 (Experimental): the observation group 2 was given Linaclotide(290 ug) in 1 day combined with 4L of Compound Polyethylene Glycol Electrolyte Powder to clear the intestine
  Interventions: Drug: Linaclotide; Drug: Compound Polyethylene Glycol Electrolyte Powder
- the observation group 3 (Experimental): the observation group 3 was given Linaclotide(290 ug) in 3 day combined with 3L of Compound Polyethylene Glycol Electrolyte Powder to clear the intestine.
  Interventions: Drug: Linaclotide; Drug: Compound Polyethylene Glycol Electrolyte Powder

INTERVENTIONS:
Drug: Linaclotide — The observation group 1 was given Linaclotide in 1 day combined with 4L of Compound Polyethylene Glycol Electrolyte Powder to clear the intestine, and the observation group 2 was given Linaclotide in 1 day combined with 4L of Compound Polyethylene Glycol Electrolyte Powder to clear the intestine. observation group 3 was given Linaclotide in 3 day combined with 3L of Compound Polyethylene Glycol Electrolyte Powder to clear the intestine. Intestinal cleanliness and the incidence of adverse reactions of patients in each group were compared.
  Arms: the observation group 1; the observation group 2; the observation group 3
Drug: Compound Polyethylene Glycol Electrolyte Powder — The control group was given Compound Polyethylene Glycol Electrolyte Powder to clear the intestines,

SUMMARY:
Constipation is a common reason of poor bowel preparation, which negatively influences the quality of colonoscopy. Clinically to explore more effective and tolerant bowel clearance programs is necessary for patients with chronic constipation.

DETAILED DESCRIPTION:
Colonoscopy is an important method to screen, diagnose and treat colon lesions. The quality of bowel preparation is requisite for the accuracy of diagnosis and safety of treatment. To explore the application effect and safety of Linaclotide combined with Compound Polyethylene Glycol Electrolyte Powder on colon cleansing before colonoscopy in patients with chronic constipation. A prospective mult-centers, colonoscopist-blinded study was conducted. A total of 300 patients with constipation who underwent colonoscopy in 8 hospitals from July to December 2021 were selected as study subjects and divided into the control group, observation group 1, observation group 2 and observation group 3 by random number table method, with 75 cases in each group. Intestinal cleanliness and the incidence of adverse reactions of patients in each group were compared.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included: The inclusion criteria were patients ≥18 years old suffering from≥2 of the following criteria of chronic constipation under the Rome IV standard: straining, hard stool, residual stool feeling, occlusion feeling, manual bowel movement(BM) performed ≥25% of overall BMs, and BM frequency<3 times a week . A chronic status was defined as symptoms being present for at least six months, with the symptoms described above being present for at least three months.

Exclusion Criteria:

* Exclusion criteria included: (1)age <18 or> 75; (2) severe chronic renal failure, severe congestive heart failure and Liver dysfunction ;(3)with uncontrolled hypertension, diabetes, intestinal obstruction, intestinal perforation and electrolyte disorders, inflammatory intestinal disease and other organic gastrointestinal diseases;(4)with neurologic, endocrine, or metabolic disorders;(5)treatment with other gastrointestinal drivers, laxatives, and antilaxatives within nearly 2 weeks;(6)history of colorectal surgery;(7) dysphagia; (8) compromised swallowing reflex or mental status;(9)with consciousness disorders or examination intolerance;(10)pregnancy or lactation;(11)allergic to the drug composition;(12)Suspected history of alcohol or substance abuse; (13)Recent participants in clinical trials; (14) unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The Boston Bowel Preparation Scale | colonoscopy screening procedure
  the effect of colon cleansing

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang L, Zhang Y, Li J, Ran Y, Wang X, Ma X, Yang Q, Wang F, Hu J, Zhuang K, Wang J, Quan X, Wang S, Meng R, Chen Y, Li X, Song Y, Han S, Hu H, Li L, Dai F. Efficacy of Polyethylene Glycol Electrolyte Powder Combined With Linaclotide for Colon Cleansing in Patients With Chronic Constipation Undergoing Colonoscopy: A Multicenter, Single-Blinded, Randomized Controlled Trial. Clin Transl Gastroenterol. 2024 Jun 1;15(6):e1. doi: 10.14309/ctg.0000000000000708. PMID 38713137